CLINICAL TRIAL: NCT05257811
Title: Earbud Electrode Electroencephalography System - Initial Feasibility Study
Brief Title: Earbud EEG Feasibility Study
Acronym: PRIME
Status: Completed | Type: Observational
Sponsor: NextSense, Inc. (Industry)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00090515
Record Dates: First submitted 2022-02-05; First posted 2022-02-25 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Epilepsy; Seizure; Sleep
Keywords: electroencephalography; polysomnography
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: NextSense EEG-enabled earbuds — Each NextSense EEGBud device includes custom-fit earbuds with biometric sensors to detect EEG, motion (via tri-axial accelerometers), and heart rate. A ring laser scanner is used to capture the unique geometry of each participant's ear and external auditory canal. Digital models of the individual ear scans are generated and used to create custom fit, 3D-printed earbuds. This design process allows for consistent contact with the inner surface of the ear canal, providing high quality signal capture of brain activity, cardiac activity, and eye movements.

SUMMARY:
The goal of this study is to characterize the ability of the NextSense ear-EEG device to detect pathologic electrographic signatures of epilepsy and physiologic signatures of sleep in subjects undergoing simultaneous inpatient continuous EEG monitoring, polysomnography, or ambulatory EEG monitoring at home.

DETAILED DESCRIPTION:
For nearly half a century, conventional electroencephalography (EEG) has been the standard of care for monitoring cerebral activity, particularly in the clinical domains of epilepsy and sleep disorders. Standard EEG involves highly time, labor, and cost intensive processes and typically requires subjects to be monitored by specially trained staff in the inpatient setting. Existing ambulatory EEG options are limited to about 3 days in duration because of decline in electrode fidelity beyond that timeframe. There is a need for unobtrusive, easy to use, longitudinal monitoring solutions that can extend to the ambulatory setting.

This study will assess whether novel NextSense EEG Earbuds are able to 1) detect seizures of varying types/localizations as well as interictal epileptiform activity (IEA) waveforms compared to simultaneously recorded conventional scalp EEG, or in some cases, intracranial EEG; and 2) detect characteristic electrographic signatures of AASM defined sleep stages compared to simultaneously recorded polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years of age and older admitted to the Epilepsy Monitoring Unit at Emory University Hospital for long-term inpatient scalp or intracranial cEEG monitoring for diagnostic or pre-surgical evaluation, or patients 18 years and older admitted to the Emory Sleep Center at the Brain Health Center for polysomnography.
* To enhance the likelihood of having a sufficient number of enrolled subjects with an adequate number of seizures, investigators may identify patients more likely to have epileptic rather than non-epileptic seizures based on the medical history.
* All patients who are undergoing ambulatory EEG monitoring at home.

Exclusion Criteria:

* Inability to safely tolerate earbuds (e.g. antecedent skin breakdown, recent injury to ear).
* Subjects who cannot have all 16 non-midline scalp EEG electrodes placed, since these EEG channels are required to accurately assess the performance of the seizure detection function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 100 patients may be invited to participate in the study. These patients will have previously been referred for admission to the epilepsy monitoring unit for either diagnostic or presurgical cEEG, or for polysomnography by the neurologists/epileptologists of the Emory Neurology Department.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Ease of use and tolerability validation of EEG earbuds for patients undergoing cEEG monitoring or polysomnography. | up to 2 weeks
  Individual tolerance success will be the presence of an interpretable EEG record for at 18 hours a day, for at least three consecutive days. Overall tolerance will be a ≥ 75% ongoing participation rate, i.e. ≤ 25% study "drop-out" rate. Patients will be questioned about the reasons they felt the EEGBuds needed to be removed, in order to improve future tolerance.
Performance validation of EEG earbuds for patients undergoing cEEG monitoring or polysomnography | up to 2 weeks
  Performance validation is measured as sensitivity (true positive) rate as defined as the total number of true detections divided by the total number of seizures; and specificity (false detection rate [FDR]) as defined as 24 x number of false detections divided by the total number of EEG hours, for each test subject. Detections will be classified as "true" or "false" based on majority rule by expert reviewers (classified by ≥ 2/3 of reviewers).
  Criteria for Success:
  1. ≥ 90% of EEG segments deemed "acceptable quality" by expert reviewers
  2. Overall seizure detection sensitivity of at least 90% and a mean FDR of no more than 5 per 24 hours
  3. Overall spike detection sensitivity of at least 90% and a mean FDR of no more than 3 per hour
  4. Overall focal slowing detection sensitivity of at least 75% and a mean FDR of no more than 3 per 24 hours (focal slowing is traditionally more difficult to ascertain so criteria will be slightly less stringent)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Winkel, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No